CLINICAL TRIAL: NCT00004233
Title: A Phase II Study of PN-401, 5-FU and Leucovorin in Unresectable or Metastatic Adenocarcinoma of the Stomach
Brief Title: S9915 Triacetyluridine, Fluorouracil, and Leucovorin in Treating Patients With Unresectable, Locally Advanced, or Metastatic Cancer of the Esophagus or Stomach
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Laurence H. Baker, D.O.; Group Chair, Southwest Oncology Group
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000067477; CA32102 (Other Grant/Funding Number: National Cancer Institute cooperative agreement); S9915 (Other: SWOG)
Record Dates: First submitted 2000-01-28; First posted 2003-08-25 (Estimated); Last update posted 2011-07-25 (Estimated); Status verified 2010-05

CONDITIONS: Esophageal Cancer; Gastric Cancer
Keywords: stage III gastric cancer; stage IV gastric cancer; recurrent gastric cancer; stage III esophageal cancer; stage IV esophageal cancer; recurrent esophageal cancer; adenocarcinoma of the stomach; adenocarcinoma of the esophagus
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms; Adenocarcinoma Of Esophagus | interventions — Fluorouracil; Leucovorin; uridine triacetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 5-FU, Leucovorin and PN-401 (Experimental): PN401 is given on Days 1-3 weekly for six weeks; 5FU and leucovorin are given on Day 1 weekely for six weeks; followed by two weeks of rest. Continued in 8 week cycles until one of the criteria for removal from treatment is met.
  Interventions: Drug: fluorouracil; Drug: leucovorin calcium; Drug: triacetyluridine

INTERVENTIONS:
Drug: fluorouracil
  Other Names: 5-FU
Drug: leucovorin calcium
  Other Names: LCV; leucovorin
Drug: triacetyluridine
  Other Names: PN-401

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Chemoprotective drugs such as triacetyluridine may protect normal cells from the side effects of chemotherapy.

PURPOSE: Phase II trial to study the effectiveness of triacetyluridine, fluorouracil, and leucovorin in treating patients who have unresectable, locally advanced, or metastatic cancer of the esophagus or stomach.

DETAILED DESCRIPTION:
OBJECTIVES:

* Assess the 6-month survival rate in patients with unresectable, locally advanced or metastatic adenocarcinoma of the stomach or gastroesophageal junction treated with triacetyluridine, fluorouracil, and leucovorin calcium.
* Evaluate the qualitative and quantitative toxic effects of this regimen in these patients.

OUTLINE: This is a multicenter study.

Patients receive leucovorin calcium IV over 2 hours and fluorouracil IV over 30 minutes beginning 1 hour into leucovorin calcium infusion on days 1, 8, 15, 22, 29, and 36. Patients receive oral triacetyluridine every 8 hours on days 1-3, 8-10, 15-17, 22-24, 29-31, and 36-38 beginning 8 hours after completion of each fluorouracil infusion. Courses repeat every 8 weeks in the absence of disease progression or unacceptable toxicity.

Patients are followed every 6 months for up to 3 years.

PROJECTED ACCRUAL: A total of 53 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically proven unresectable, locally advanced or metastatic adenocarcinoma of the stomach or gastroesophageal junction
* No known brain metastases

  * Negative brain imaging required for neurologic signs and symptoms

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Zubrod 0-1

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count greater than 100,000/mm^3

Hepatic:

* Bilirubin no greater than upper limit of normal (ULN)
* SGOT or SGPT no greater than 1.5 times ULN (5 times ULN if liver tumor present)

Renal:

* Creatinine no greater than ULN

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception
* Must be able to swallow oral medication
* No AIDS syndrome or HIV-associated complex
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or adequately treated stage I or II cancer in complete remission

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior biologic therapy
* No concurrent biologic therapy

Chemotherapy:

* No prior chemotherapy for advanced or metastatic gastric cancer
* At least 6 months since prior chemotherapy as adjuvant or radiation sensitizer

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 1 month since prior radiotherapy and recovered
* No concurrent radiotherapy

Surgery:

* At least 3 weeks since prior major surgical resection of intra-abdominal organs and recovered

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2001-02; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Six month survival | six months after registration

SECONDARY OUTCOMES:
evaluate quantitative and qualitative toxicities | three years at most

CONTACTS AND LOCATIONS:
Overall Officials: James H. Doroshow, MD, Study Chair — City of Hope Comprehensive Cancer Center
Locations (97):
- United States (97):
  - MBCCOP - Gulf Coast, Mobile, Alabama
  - CCOP - Greater Phoenix, Phoenix, Arizona
  - Veterans Affairs Medical Center - Phoenix (Hayden), Phoenix, Arizona
  - Veterans Affairs Medical Center - Tucson, Tucson, Arizona
  - Arizona Cancer Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Veterans Affairs Medical Center - Little Rock (McClellan), Little Rock, Arkansas
  - Cancer Center and Beckman Research Institute, City of Hope, Duarte, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Veterans Affairs Medical Center - West Los Angeles, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Veterans Affairs Outpatient Clinic - Martinez, Martinez, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - University of California Davis Medical Center, Sacramento, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - David Grant Medical Center, Travis Air Force Base, California
  - University of Colorado Cancer Center, Denver, Colorado
  - Veterans Affairs Medical Center - Denver, Denver, Colorado
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Dwight David Eisenhower Army Medical Center, Fort Gordon, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - MBCCOP - University of Illinois at Chicago, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago (Westside Hospital), Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - Veterans Affairs Medical Center - Hines (Hines Junior VA Hospital), Hines, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Lexington, Lexington, Kentucky
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Veterans Affairs Medical Center - New Orleans, New Orleans, Louisiana
  - Louisiana State University Health Sciences Center - Shreveport, Shreveport, Louisiana
  - Veterans Affairs Medical Center - Shreveport, Shreveport, Louisiana
  - Boston Medical Center, Boston, Massachusetts
  - Veterans Affairs Medical Center - Boston (Jamaica Plain), Jamaica Plain, Massachusetts
  - Veterans Affairs Medical Center - Ann Arbor, Ann Arbor, Michigan
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Veterans Affairs Medical Center - Detroit, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - CCOP - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - Providence Hospital - Southfield, Southfield, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - Veterans Affairs Medical Center - Biloxi, Biloxi, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Veterans Affairs Medical Center - Jackson, Jackson, Mississippi
  - Keesler Medical Center - Keesler AFB, Keesler Air Force Base, Mississippi
  - Veterans Affairs Medical Center - Kansas City, Kansas City, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. Louis University Health Sciences Center, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Veterans Affairs Medical Center - Albuquerque, Albuquerque, New Mexico
  - MBCCOP - University of New Mexico HSC, Albuquerque, New Mexico
  - Veterans Affairs Medical Center - Albany, Albany, New York
  - St. Vincents Comprehensive Cancer Center, New York, New York
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Veterans Affairs Medical Center - Cincinnati, Cincinnati, Ohio
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Kettering, Ohio
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - Veterans Affairs Medical Center - Oklahoma City, Oklahoma City, Oklahoma
  - Oregon Cancer Center, Portland, Oregon
  - Veterans Affairs Medical Center - Portland, Portland, Oregon
  - CCOP - Columbia River Program, Portland, Oregon
  - Veterans Affairs Medical Center - Charleston, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Veterans Affairs Medical Center - Houston, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Veterans Affairs Medical Center - San Antonio (Murphy), San Antonio, Texas
  - Veterans Affairs Medical Center - Temple, Temple, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Veterans Affairs Medical Center - Salt Lake City, Salt Lake City, Utah
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Swedish Cancer Institute, Seattle, Washington
  - Veterans Affairs Medical Center - Seattle, Seattle, Washington
  - CCOP - Northwest, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington

REFERENCES:
- [Result] Doroshow JH, McCoy S, Macdonald JS, Issell BF, Patel T, Cobb PW, Yost KJ, Abbruzzese JL. Phase II trial of PN401, 5-FU, and leucovorin in unresectable or metastatic adenocarcinoma of the stomach: a Southwest Oncology Group study. Invest New Drugs. 2006 Nov;24(6):537-42. doi: 10.1007/s10637-006-9244-8. PMID 16832602